CLINICAL TRIAL: NCT04641104
Title: The Thiamine Administration After Cardiac Surgery Trial
Acronym: TAACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarah Saxena (Other)
Collaborators: CHU de Charleroi (Other)
Responsible Party: Sponsor-Investigator, Sarah Saxena, MD, Université Libre de Bruxelles
Organization: Université Libre de Bruxelles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAACS trial
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Lactate Blood Increase; Thiamine Deficiency
MeSH Terms: conditions — Hyperlactatemia; Thiamine Deficiency | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: This is a monocentric randomized, controlled, double blind study in patients undergoing elective cardiac surgery with extra corporal circulation. Anesthesia management of these patients is standardised in terms of volume-controlled ventilation, fluid and inotropes management.
  Randomization of 100 patients for the administration, of a solution of 500 mg of Thiamine Hydrocloride in a solution of 100 ml of NaCl 0.9% versus a solution of 100 ml of NaCl 0.9% alone in adult patients (≥ 18 years-old) with a lactate ≥ 2 mmol / L in the first 6 hours of ICU admission.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiamine (Experimental): Patients in this arm will receive a solution of 500 mg of Thiamine Hydrocloride in a solution of 100 ml of NaCl 0.9%.
  Interventions: Drug: Thiamine 500 MG
- Placebo (Placebo Comparator): Patients in this arm will receive a solution of 100 ml of NaCl 0.9% alone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiamine 500 MG — A solution of 500 mg of Thiamine Hydrocloride in a solution of 100 ml of NaCl 0.9% will be administered post-cardiac surgery in patients with lactate levels ≥ 2 mmol / L in the first 6 hours post-ICU admission.
  Other Names: Thiamine
  Arms: Thiamine
Drug: Placebo — 100 ml of NaCl 0.9% will be administered in the placebo group.
  Arms: Placebo

SUMMARY:
Thiamine (Vitamin B1) is essential for cell function and as a co-factor of the enzyme Pyruvate Dehydrogenase to initiate the Krebs cycle and thus the aerobic metabolism of glucose.

We hypothesize that thiamine supplementation improves the clearance of lactate in the first 24 hours after cardiac surgery with extracorporeal circulation in patients with high lactate concentration.

DETAILED DESCRIPTION:
Thiamine (Vitamin B1) is essential for cell function and as a co-factor of the enzyme Pyruvate Dehydrogenase to initiate the Krebs cycle and thus the aerobic metabolism of glucose.

Thiamine deficiency, can be caused by alcoholism or bariatric surgery and is associated with severe complications such as Wernicke's encephalopathy or Beri-Beri syndrome.

Thiamine deficiency can also be the cause for an increase in lactate levels due to the transformation of pyruvate to lactate. An increase in lactate levels is associated with a worse prognostic. A decrease is, on the contrary, associated with an improved prognostic, during CPR and also after cardiac arrest.

Recently, studies have shown that thiamine deficiency is underdiagnosed in ICU patients.

On top of this, extra-corporeal circulation can worsen this deficiency. This could explain why certain on-pump cardiac surgery patients have increased lactate levels post-operatively, despite optimal blood pressure, cardiac output, diuresis, peripheral perfusion Donnino et al have shown that in a sepsis context thiamine administration improved lactate clearance during the first 24 hours of ICU admission and improved mortality rates at 28 days post-ICU admission.

Therefore, the hypothesis of this study is that thiamine supplementation improves the clearance of lactate in the first 24 hours after cardiac surgery with extracorporeal circulation in patients with high lactate concentration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective cardiac surgery with extra-corporeal circulation in the CHU de Charleroi between November 2020 and December 2021. Written informed consent will be obtained from each patient/ family member participating in the study.

Exclusion Criteria:

* Patients already supplemented with vitamins
* Patients with an allergy to thiamine
* Patients who are priorly treated with linezolide, antiretrovirals and/or metformin treatment within 48 hours preoperatively
* Patients with mitochondrial disorders
* Patients with Child Pugh C cirrhosis
* Patients with a history of epilepsy with tonic-clonic movements postoperatively.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Lactate | 24 hours
  Lactate level will be specifically be measured 24h post-ICU admission to evaluate the effect of thiamine versus placebo.

SECONDARY OUTCOMES:
Fluid balance | 48 hours
  The influence of thiamine/placebo on the use of volume expansion during ICU stay will also be evaluated
Inotropes | 48 hours
  The influence of thiamine: placebo on the use of inotropes during ICU stay will also be evaluated
Mechanical ventilation | 48 hours
  The influence of thiamine/ placebo on extubation time will also be evaluated.
Length of ICU stay | 5 days
  The influence of thiamine/ placebo on ICU discharge will also be evaluated.
Length of hospital stay | 30 days
  The influence of thiamine/ placebo on hospital discharge will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: MIchael Piagnerelli, MD; PHD, Principal Investigator — CHU de Charleroi, Belgium
Locations (1):
- CHU-Charleroi Hopital Civil Marie Curie, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frank RA, Leeper FJ, Luisi BF. Structure, mechanism and catalytic duality of thiamine-dependent enzymes. Cell Mol Life Sci. 2007 Apr;64(7-8):892-905. doi: 10.1007/s00018-007-6423-5. PMID 17429582
- [Result] Collie JTB, Greaves RF, Jones OAH, Lam Q, Eastwood GM, Bellomo R. Vitamin B1 in critically ill patients: needs and challenges. Clin Chem Lab Med. 2017 Oct 26;55(11):1652-1668. doi: 10.1515/cclm-2017-0054. PMID 28432843
- [Result] Flannery AH, Adkins DA, Cook AM. Unpeeling the Evidence for the Banana Bag: Evidence-Based Recommendations for the Management of Alcohol-Associated Vitamin and Electrolyte Deficiencies in the ICU. Crit Care Med. 2016 Aug;44(8):1545-52. doi: 10.1097/CCM.0000000000001659. PMID 27002274
- [Result] Nichol AD, Egi M, Pettila V, Bellomo R, French C, Hart G, Davies A, Stachowski E, Reade MC, Bailey M, Cooper DJ. Relative hyperlactatemia and hospital mortality in critically ill patients: a retrospective multi-centre study. Crit Care. 2010;14(1):R25. doi: 10.1186/cc8888. Epub 2010 Feb 24. PMID 20181242
- [Result] Mikkelsen ME, Miltiades AN, Gaieski DF, Goyal M, Fuchs BD, Shah CV, Bellamy SL, Christie JD. Serum lactate is associated with mortality in severe sepsis independent of organ failure and shock. Crit Care Med. 2009 May;37(5):1670-7. doi: 10.1097/CCM.0b013e31819fcf68. PMID 19325467
- [Result] Sterling SA, Puskarich MA, Shapiro NI, Trzeciak S, Kline JA, Summers RL, Jones AE; Emergency Medicine Shock Research Network (EMSHOCKNET). Characteristics and outcomes of patients with vasoplegic versus tissue dysoxic septic shock. Shock. 2013 Jul;40(1):11-4. doi: 10.1097/SHK.0b013e318298836d. PMID 23649098
- [Result] Casserly B, Phillips GS, Schorr C, Dellinger RP, Townsend SR, Osborn TM, Reinhart K, Selvakumar N, Levy MM. Lactate measurements in sepsis-induced tissue hypoperfusion: results from the Surviving Sepsis Campaign database. Crit Care Med. 2015 Mar;43(3):567-73. doi: 10.1097/CCM.0000000000000742. PMID 25479113
- [Result] Vellinga NAR, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, van der Voort PHJ, Dondorp AM, Bafi T, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Bakker J, Ince C; microSOAP study group. Mildly elevated lactate levels are associated with microcirculatory flow abnormalities and increased mortality: a microSOAP post hoc analysis. Crit Care. 2017 Oct 18;21(1):255. doi: 10.1186/s13054-017-1842-7. PMID 29047411
- [Result] Nguyen HB, Rivers EP, Knoblich BP, Jacobsen G, Muzzin A, Ressler JA, Tomlanovich MC. Early lactate clearance is associated with improved outcome in severe sepsis and septic shock. Crit Care Med. 2004 Aug;32(8):1637-42. doi: 10.1097/01.ccm.0000132904.35713.a7. PMID 15286537
- [Result] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Result] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176
- [Result] Pan J, Peng M, Liao C, Hu X, Wang A, Li X. Relative efficacy and safety of early lactate clearance-guided therapy resuscitation in patients with sepsis: A meta-analysis. Medicine (Baltimore). 2019 Feb;98(8):e14453. doi: 10.1097/MD.0000000000014453. PMID 30813144
- [Result] Donnino MW, Miller J, Goyal N, Loomba M, Sankey SS, Dolcourt B, Sherwin R, Otero R, Wira C. Effective lactate clearance is associated with improved outcome in post-cardiac arrest patients. Resuscitation. 2007 Nov;75(2):229-34. doi: 10.1016/j.resuscitation.2007.03.021. Epub 2007 Jun 20. PMID 17583412
- [Result] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Result] Costa NA, Gut AL, de Souza Dorna M, Pimentel JA, Cozzolino SM, Azevedo PS, Fernandes AA, Zornoff LA, de Paiva SA, Minicucci MF. Serum thiamine concentration and oxidative stress as predictors of mortality in patients with septic shock. J Crit Care. 2014 Apr;29(2):249-52. doi: 10.1016/j.jcrc.2013.12.004. Epub 2013 Dec 14. PMID 24412011
- [Result] Donnino MW, Carney E, Cocchi MN, Barbash I, Chase M, Joyce N, Chou PP, Ngo L. Thiamine deficiency in critically ill patients with sepsis. J Crit Care. 2010 Dec;25(4):576-81. doi: 10.1016/j.jcrc.2010.03.003. Epub 2010 Jun 19. PMID 20646908